CLINICAL TRIAL: NCT01737918
Title: Phase 1/2 Study of the Effect of TOT or Solifenacin After Cesa or Vasa on Urge Urinary Incontinence
Brief Title: Treatment of Urge Urinary Incontinence in Women After Failure of Cesa or Vasa
Acronym: URGE-II
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Klinikum der Universität Köln (Other)
Responsible Party: Principal Investigator, Professor Dr. Wolfram Jäger, Professor, Klinikum der Universität Köln
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: URGE-II
Record Dates: First submitted 2012-11-28; First posted 2012-11-30 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Surgical Treatment of Urge Incontinence
Keywords: urge urinary incontinence, cesa, vasa, TOT, solifenacin
MeSH Terms: conditions — Urinary Incontinence, Urge | interventions — Solifenacin Succinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- trans obturatorial tape (TOT) (Experimental): placement of a sub-urethral tape
  Interventions: Procedure: TOT
- solifenacin (Active Comparator): 10 mg per day
  Interventions: Drug: solifenacin

INTERVENTIONS:
Procedure: TOT
  Other Names: trans obturatorial tape
  Arms: trans obturatorial tape (TOT)
Drug: solifenacin
  Other Names: VESICUR 10mg per day
  Arms: solifenacin

SUMMARY:
Urge urinary incontinence can be a disorder caused by destroyed pelvic structures. We repaired the uteri-sacral ligaments (USL) by cesa or vasa. The study evaluates if solifenacin can lead to continence after surgery or if also the pubo-urethral ligaments (PUL) need to be repaired.

DETAILED DESCRIPTION:
It was hypothesized that urge urinary incontinence in women is based on the destruction of the uteri-sacral ligaments (USL)and the pubourethral ligaments (PUL). In a preliminary study (URGE I) we repaired the USL by cesa or vasa. Those patients who are still incontinent after cesa and vasa get the repair of the PUL by means of trans-obturator tapes (TOT). That treatment is compared to conservative medical treatment. Cross over after completion of three months is possible if no continence is achieved.

ELIGIBILITY:
Inclusion Criteria:

* prior vasa or cesa operation as part of the URGE I study
* stress urinary incontinence
* mixed urinary incontinence

Exclusion Criteria:

* previous urogynecological surgery
* avulsion of cesa or vasa tape
* pregnancy
* neurologic/psychological reasons for incontinence
* body weight >100kg
* syndrome of dry overactive bladder

Ages: 40 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2013-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
cure of incontinence | 3 months

SECONDARY OUTCOMES:
improvement of urge symptoms | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Wolfram H Jager, PhD, Principal Investigator — Study Supervisor
Locations (1):
- Abt. Beckenbodenchirurgie der Universitäts-Frauenklinik Köln, Cologne, North Rhine-Westphalia, Germany